CLINICAL TRIAL: NCT00901121
Title: Maxillary Sinus Grafting With Bio-Oss or Straumann Bone Ceramic Followed by Delayed Placement of Straumann Dental Implants: A Comparative Histomorphometric and Clinical Study
Brief Title: Maxillary Sinus Elevation With Bio-Oss or Straumann BoneCeramic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 09/04
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Teeth Loss; Bone Loss
Keywords: maxillary sinus lift; Histomorphometric evaluation; bone graft; bone augmentation
MeSH Terms: conditions — Anodontia; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BoneCeramic (Experimental): Straumann BoneCeramic is a fully synthetic bone graft substitute of medical grade purity in particulate form composed of biphasic calcium phosphate - a mixture of 60% hydroxylapatite and of 40% of the beta form of tricalcium phosphate (beta-TCP).
  Interventions: Device: Straumann BoneCeramic
- Bio-Oss (Active Comparator): Bio-Oss spongiosa granules, size of particle 0.25-1 mm
  Interventions: Device: Bio-Oss

INTERVENTIONS:
Device: Straumann BoneCeramic — Straumann BoneCeramic (500-1000 microns, 0.5g)
  Arms: BoneCeramic
Device: Bio-Oss — Bio-Oss spongiosa granules, size of particle 0.25-1 mm
  Arms: Bio-Oss

SUMMARY:
The purpose of the study was to test a clinically relevant non-inferiority of Straumann BoneCeramic treatment compared to Bio-Oss treatment 180 to 240 days after sinus grafting procedure.

DETAILED DESCRIPTION:
This is a prospective, controlled, randomised, multicenter study. The total study duration for each patient should be three years.

In total 13 visits per patient are scheduled in this study.

The study device Straumann Bone Ceramic is CE-marked.

Height centers in Italy will participate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females were at least 18 years of age and not more than 70 years old
* A dental implant procedure was foreseen in the maxilla region corresponding to maxillary sinus
* Patients presented a bone defect in the sinus area, which needed a sinus floor elevation to place one or more dental implants
* The patients were unilaterally or bilaterally edentulous in the maxillary region corresponding to the sinuses
* Residual alveolar crest height of the lateral-posterior segments of the edentulous maxilla below the floor of the maxillary sinus was less than 8 mm and at least 3 mm, measured by CT scans. Furthermore, residual alveolar crest width should be at least in average 6 mm measured by the CT scans
* Patients were committed to the study
* Patients were healthy at time of surgery

Exclusion Criteria:

* Medical conditions requiring prolonged use of steroids
* Standard blood test performed by the medical practitioner of the patient showing: leukocyte dysfunction and deficiencies
* Haemophilia, bleeding disorders or cumarin therapy
* History of neoplastic disease requiring the use of chemotherapy
* History of radiation therapy to the head and neck
* Patients with history of renal failure or chronic renal diseases
* Patients affected by chronic liver diseases
* Patients with severe or uncontrolled metabolic bone disorders
* Uncontrolled endocrine disorders (including diabetes)
* Current pregnancy at the time of recruitment
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 90 days period immediately prior to implant surgery on study day 0
* Alcoholism or chronically drug abuse causing systemic compromisation
* Immunocompromised patients including patients infected with HIV
* Patients who smoke more than 10 cigarettes per day or cigar equivalents, or who chew tobacco
* Conditions or circumstances, in the opinion of the investigator, which could represent a general contra-indication for surgical procedure or would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability

Local exclusion criteria

* Local inflammation, including untreated periodontitis to residual dentition
* Mucosal diseases such as erosive lichen planus
* History of local radiation therapy
* Presence of oral lesions (such as ulceration, malignancy)
* Severe bruxing or clenching habits
* Persistent intraoral infection
* Patients with inadequate oral hygiene or unmotivated for adequate home care
* Unhealed extraction sites in the upper premolar or molar area
* Last tooth extraction performed less than 3 months before surgery 1
* Previous GBR (guided bone regeneration) or dental implant treatment in the lateral-posterior segments of the upper maxilla (foreseen implant site)
* Patients presenting clinical and radiological signs and symptoms of maxillary sinus disease
* Patients presenting with residual alveolar crest height of the lateral-posterior segments of the edentulous maxilla below the floor of the maxillary sinus less than 3 mm and residual alveolar crest width less than 6 mm (measured by the CT scans)
* The reduction in residual bone height was determined by sinus pneumatization and not by vertical resorption of the residual alveolar crest with increased interarch distance. Patients with increased interarch distance were excluded from the study
* Existing teeth in the residual dentition with untreated endodontic or cariologic problems
* Horizontal or vertical augmentation to correct the vertical inter-arch distance or to correct horizontal defects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-07; Primary Completion 2007-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Histological evaluation of the ratio between new bone and residual graft material at the implant site 180 to 240 days after graft-placement. | 180 to 240 days

SECONDARY OUTCOMES:
Histomorphometric evaluation of the amount of new bone, soft tissue and remaining graft in the treatment, control and in a 1mm compartment 1mm close to the autogenous bone and the amount of new bone on contact with the graft. | 180 to 240 days
Evaluation of the survival and success rate of Straumann dental implants placed in the grafted areas | 3 years
Clinical evaluation of peri implant soft tissue | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Chiapasco, Prof, Principal Investigator — University of Milan
Locations (6):
- Italy (6):
  - Private Practice, Milan
  - University of Milan, Milan
  - Private Practice, Naples
  - Private Practice, Pavia
  - Private Practice, Rome
  - Eastman Dental Hospital ASL RMA Roma, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cordaro L, Bosshardt DD, Palattella P, Rao W, Serino G, Chiapasco M. Maxillary sinus grafting with Bio-Oss or Straumann Bone Ceramic: histomorphometric results from a randomized controlled multicenter clinical trial. Clin Oral Implants Res. 2008 Aug;19(8):796-803. doi: 10.1111/j.1600-0501.2008.01565.x. PMID 18705811